CLINICAL TRIAL: NCT07361874
Title: IMPACT-MACS Study: Investigating the Mechanisms, Pathophysiology, and Cardiometabolic Treatment in Mild Autonomous Cortisol Secretion
Brief Title: IMPACT-MACS: Adrenalectomy vs Semaglutide for Metabolic Outcomes in Mild Autonomous Cortisol Secretion
Acronym: IMPACT-MACS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Oksana Hamidi, DO, MSCS, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU20251717; 1K23DK142038-01A1 (NIH)
Record Dates: First submitted 2026-01-20; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Mild Autonomous Cortisol Secretion (MACS); Autonomous Cortisol Secretion (ACS); Subclinical Cushing's; Mild Autonomous Cortisol Excess
Keywords: Mild Autonomous Cortisol Secretion; MACS; Adrenal incidentaloma; Adrenal adenoma; Subclinical Cushing; Hypercortisolism; Cortisol dysregulation; Adrenalectomy; Semaglutide; Weight loss; Body composition; Insulin resistance; GLP-1 receptor agonist; Hyperinsulinemic-euglycemic clamp; Cortisol dynamics; Visceral fat; cardiometabolic risk; randomized controlled trial
MeSH Terms: conditions — Adrenal incidentaloma; ACTH Syndrome, Ectopic; Cushing Syndrome; Weight Loss; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: This study includes two coordinated components. First, a randomized controlled trial in adults with mild autonomous cortisol secretion (MACS) who are eligible for adrenalectomy. Participants are randomized 1:1 to adrenalectomy or semaglutide for 26 weeks, stratified by post-DST cortisol and sex. This evaluates surgical versus medical effects on insulin sensitivity and cortisol regulation.
  Second, a matched case-control comparison in adults without adrenal tumors who receive semaglutide using the same schedule. Controls are matched 1:1 by age, sex, BMI, and diabetes status to isolate disease-specific metabolic responses.
  Both components follow identical assessments in an open-label, parallel-assignment design without crossover, enabling evaluation of treatment modality in MACS and differential response to semaglutide.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Adrenalectomy (MACS) (Active Comparator): Adults with mild autonomous cortisol secretion (MACS) who are clinically eligible for adrenalectomy undergo unilateral adrenalectomy as part of standard care. Participants complete all metabolic assessments before and after treatment.
  Interventions: Procedure: Intervention 1: Adrenalectomy
- Arm 2: Semaglutide (MACS) (Active Comparator): Adults with MACS receive once-weekly semaglutide for 26 weeks using FDA-approved weight-management dosing. Participants undergo the same assessments as the surgery group.
  Interventions: Drug: Intervention 2: Semaglutide
- Arm 3: Semaglutide (Matched Controls) (Active Comparator): Matched adults without adrenal tumors receive semaglutide using the same dosing schedule as MACS participants. This arm allows comparison of semaglutide responses between individuals with and without cortisol dysregulation.
  Interventions: Drug: Intervention 2: Semaglutide

INTERVENTIONS:
Procedure: Intervention 1: Adrenalectomy — Surgical removal of one adrenal gland performed by an endocrine surgeon following institutional standard-of-care practices. Includes postoperative monitoring for adrenal insufficiency and routine clinical follow-up.
  Arms: Arm 1: Adrenalectomy (MACS)
Drug: Intervention 2: Semaglutide — Once-weekly subcutaneous semaglutide administered according to FDA-approved titration for chronic weight management (0.25 mg to 2.4 mg weekly as tolerated). Participants receive training on injection technique, dose escalation, and safety monitoring.
  Arms: Arm 2: Semaglutide (MACS); Arm 3: Semaglutide (Matched Controls)

SUMMARY:
The goal of this study is to learn how two treatments-adrenalectomy (surgical removal of an adrenal gland) and semaglutide (a medication used for weight management)-affect insulin resistance and cortisol regulation in adults with mild autonomous cortisol secretion (MACS). The study will also learn how these treatments impact body composition, blood pressure, cholesterol, inflammation, muscle strength, and quality of life.

The main questions the study aims to answer are:

1. Does adrenalectomy or semaglutide improve insulin resistance more in people with MACS?
2. How do these treatments change cortisol patterns and other cardiometabolic risk factors?
3. Do people with MACS respond differently to semaglutide compared to matched adults without MACS?

Participants will:

1. Receive either adrenalectomy or semaglutide if they have MACS, or semaglutide if they are matched controls
2. Complete clinic visits and phone visits over about 26-30 weeks
3. Undergo metabolic testing such as blood tests, urine steroid profiling, body composition scans, blood pressure monitoring, muscle strength testing, and questionnaires about health and well-being

DETAILED DESCRIPTION:
This single-center, prospective, interventional study evaluates metabolic responses to surgical versus medical treatment in adults with mild autonomous cortisol secretion (MACS). The study includes:

1. a randomized controlled trial comparing adrenalectomy to semaglutide in MACS, and
2. a parallel matched case-control comparison evaluating semaglutide effects in MACS versus matched controls without adrenal tumors.

The primary objective is to compare changes in insulin sensitivity measured by hyperinsulinemic-euglycemic clamp (M-value) from baseline to week 26. Secondary outcomes include cortisol dynamics, steroid profiling, cardiometabolic biomarkers, body composition, blood pressure, muscle strength, and patient-reported quality of life.

Semaglutide is administered within its FDA-approved indication for weight management; adrenalectomy is standard of care. No investigational drugs or devices are used, and no IND is required.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years
* MACS groups: adrenal adenoma + DST cortisol >1.8 µg/dL + no overt Cushing + eligible for adrenalectomy
* Willingness to postpone surgery 6 months if randomized
* Controls: no adrenal abnormalities + normal DST + BMI ≥27 + ≥2 cardiometabolic conditions
* Stable medication doses for ≥4 weeks
* Negative pregnancy test if applicable

Exclusion Criteria:

* Prior GLP-1 RA within 90 days
* Weight change >5 kg in past 90 days
* Prior obesity/diabetes surgery
* Type 1 diabetes or other diabetes types
* Severe organ disease
* Recent pancreatitis
* Pregnancy, breastfeeding
* Contraindication to semaglutide
* Contraindication to surgery delay
* Chronic glucocorticoid use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2030-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Insulin Sensitivity (M-value), mg/kg/min | Baseline to Week 26
  Hyperinsulinemic-euglycemic clamp

SECONDARY OUTCOMES:
Change in fasting plasma glucose, mg/dL | Baseline to Week 26
Change in hemoglobin A1C, % | Baseline to Week 26
  fasting blood test
Change in fasting insulin, µU/mL | Baseline to Week 26
  Fasting blood test
Change in glucagon, pg/mL | Baseline to Week 26
  Fasting blood test
Change in c-peptide, nmol/L | Baseline to Week 26
  Fasting blood test
Change in IGF-1, ng/mL | Baseline to Week 26
  Fasting blood glucose
Change in IGF-II, ng/mL | Baseline to Week 26
  Fasting blood test
Change in IGFBP-1, ng/mL | Baseline to Week 26
  Fasting blood test
Change in leptin, ng/mL | Baseline to Week 26
  Fasting blood glucose
Change in adiponectin, μg/mL | Baseline to Week 26
  Fasting blood test
% of patients with normal dexamethasone suppression test, % | Baseline to Week 26
  1-mg dexamethasone suppression test
Change in steroid profile, ng/24h | Baseline to Week 26
  25-steroid profiling in the 24-hour urine, reported as aggregate
Mean change in systolic BP, mmHg | Baseline to Week 26
  24-hour Ambulatory BP
Mean change in diastolic BP, mmHg | Baseline to Week 26
  24-hour Ambulatory BP
Change in cholesterol, mg/dL | Baseline to Week 26
  Fasting blood test
Change in Free Fatty Acids, mmol/L | Baseline to Week 26Baseline to Week 26
  Fasting blood test
Change in C-reactive protein, pg/mL | Baseline to Week 26
  Fasting blood test
Change in TNF-alpha, pg/mL | Baseline to Week 26
  Fasting blood glucose
Change in Interleukin-1, pg/mL | Baseline to Week 26
  Fasting blood test
Change in Interleukin-6, pg/mL | Baseline to Week 26
  Fasting blood test
Change in body weight, kg | Baseline to Week 26
  electronic scale
Change in BMI, kg/m2 | Baseline to Week 26
  calculated from weight and height
Change in waist circumference, cm | Baseline to Week 26
  Tape measure
Change in fat area, cm2 | Baseline to Week 26
  Limited unenhanced CT
Change in muscle area, cm2 | Baseline to Week 26
  Limited unenhanced CT
Change in bone mineral density, mg/cm³ | Baseline to Week 26
  Limited unenhanced CT
Change in chair rise test, stands/30s | Baseline to Week 26
  Time test, number of stands from chair in 30 seconds
Change in Hand Grip Strength, kg | Baseline to Week 26
  Dynamometer
Change in overall quality of life, score | Baseline to Week 26
  PROMIS Global Health Questionnaire, domain-specific scales;
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health v1.2 Questionnaire assesses overall health-related quality of life across multiple domains, including physical health, mental health, social functioning, fatigue, and general well-being. It yields two standardized T-score summary measures (Global Physical Health and Global Mental Health).
  Score Range: T-scores typically range from 20 to 80. Interpretation: Higher T-scores indicate better health-related quality of life. Assessment Method: Self-report questionnaire; estimated completion time 2-5 minutes.
Change in disease-specific QoL, score | Baseline to Week 26
  Cushing Quality of Life Questionnaire (CushingQoL)
  Description:
  The Cushing Quality of Life Questionnaire (CushingQoL) is a disease-specific tool assessing health-related quality of life in individuals with hypercortisolism. It contains 12 items scored on a 5-point Likert scale.
  Score Range: 12 (minimum) to 60 (maximum). Interpretation: Higher scores indicate better quality of life; lower scores indicate poorer quality of life.
  Domains: Sleep disturbances, mood, physical appearance, social interaction, health concerns.
  Assessment Method: Self-administered; estimated completion time ~5 minutes.
Change in mood, score | Baseline to Week 26
  PROMIS Depression Short Form & PROMIS Anxiety Short Form
  Description:
  The PROMIS Depression Short Form and PROMIS Anxiety Short Form measure depressive and anxiety symptoms over the past seven days, assessing emotional distress, negative affect, and somatic symptoms. Responses are on a 5-point Likert scale ("Never" to "Always"), converted to standardized T-scores.
  Score Range: T-scores typically range from 20 to 80. Interpretation: Higher scores indicate worse depressive or anxiety symptoms. Assessment Method: Self-report questionnaires; estimated completion time 2-4 minutes each.
Change in cognition, seconds | Baseline to Week 26
  Trail Making Test - Part A and Part B (TMT-A and TMT-B)
  Description:
  The Trail Making Test Parts A and B assess visual attention, processing speed, cognitive flexibility, and executive function. Part A requires sequential connection of numbers; Part B requires alternating between numbers and letters.
  Score Range: 0 to 300 seconds (maximum test time). Interpretation: Higher (longer) completion times indicate worse cognitive performance.
  Assessment Method: Performance-based timed test administered by study personnel; expected duration ~5 minutes.
Change in sleep, score | Baseline to Week 26
  PROMIS Sleep Disturbance Short Form
  Description:
  The PROMIS Sleep Disturbance Short Form evaluates sleep quality, difficulty initiating and maintaining sleep, and overall sleep problems over the past seven days. Scores are converted into standardized T-scores.
  Score Range: T-scores typically range from 20 to 80. Interpretation: Higher scores indicate worse sleep disturbance. Assessment Method: Self-administered; estimated completion time 2-4 minutes.
Change in frailty, score | Baseline to Week 26
  FRAIL Scale (Fatigue, Resistance, Ambulation, Illnesses, Loss of Weight)
  Description:
  The FRAIL Scale is a validated screening instrument assessing functional decline and physiological frailty. It consists of five yes/no items: fatigue, resistance, ambulation, illnesses, and weight loss.
  Score Range: 0 (minimum) to 5 (maximum). Interpretation: Higher scores indicate greater frailty.
  Frailty Categories:
  0: Robust 1-2: Pre-frail 3-5: Frail
  Assessment Method: Administered by study personnel; duration ~1 minute.
Change in eating behavior, score | Baseline to Week 26
  Eating Behavior and Appetite Questionnaire (EBAQ)
  Description:
  The Eating Behavior and Appetite Questionnaire (EBAQ) evaluates hunger, satiety, food cravings, and changes in appetite and eating behavior. It generates domain-specific and total scores.
  Score Range: Varies by version; treated as continuous scores with defined minimum and maximum values per subscale.
  Interpretation: Higher scores indicate greater appetite or more pronounced eating-behavior disturbances.
  Assessment Method: Self-administered; estimated completion time 3-5 minutes.
Adverse Events and Serious Adverse Events | Baseline through Week 30

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) from the IMPACT-MACS study will be shared in accordance with NIH Data Management and Sharing Policy. Shared IPD will include primary and secondary outcome data such as insulin sensitivity (M-value), hormonal and cardiometabolic biomarkers, body composition measures, ambulatory blood pressure data, physical function tests, patient-reported outcomes, and adverse events. No genetic data will be shared. IPD will become available at the time of primary publication or by the end of the award period, expected by Q2 2030. Data will be accessible to qualified investigators for biomedical research through the NIDDK Central Repository, with requests managed under a Data Use Agreement. IRB approval or exemption is required, and data may not be used for ancestry or non-biomedical research.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Start Date:
  Individual participant data (IPD) and supporting documents will become available at the time of primary results publication or by the end of the study award period, whichever occurs first. Availability is expected to begin by Q2 2030.
  End Date:
  IPD will remain available indefinitely through the NIDDK Central Repository, as long as the repository remains active and able to distribute the data under its Data Use Agreement procedures.
Access Criteria: Individual participant data (IPD) and supporting materials will be available to qualified investigators conducting health-related, medical, or biomedical research. Requestors must submit a research proposal and obtain institutional IRB approval or exemption before access is granted.
  Data will be shared in de-identified form through the NIDDK Central Repository, which manages requests under its governed Data Use Agreement (DUA) process. Approved investigators will be able to access the de-identified IPD, study protocol, and data dictionary through the repository's secure system. No identifiable information or genetic data will be shared.
URL: https://reporter.nih.gov/search/14E9CE024F8FC3D67598B8961CAA4A01A2FFCEB861BF/project-details/11230185#similar-Projects

REFERENCES:
- [Background] Yozamp N, Vaidya A. Assessment of mild autonomous cortisol secretion among incidentally discovered adrenal masses. Best Pract Res Clin Endocrinol Metab. 2021 Jan;35(1):101491. doi: 10.1016/j.beem.2021.101491. Epub 2021 Feb 6. PMID 33593680
- [Background] Bancos I, Prete A. Approach to the Patient With Adrenal Incidentaloma. J Clin Endocrinol Metab. 2021 Oct 21;106(11):3331-3353. doi: 10.1210/clinem/dgab512. PMID 34260734
- [Background] Prete A, Subramanian A, Bancos I, Chortis V, Tsagarakis S, Lang K, Macech M, Delivanis DA, Pupovac ID, Reimondo G, Marina LV, Deutschbein T, Balomenaki M, O'Reilly MW, Gilligan LC, Jenkinson C, Bednarczuk T, Zhang CD, Dusek T, Diamantopoulos A, Asia M, Kondracka A, Li D, Masjkur JR, Quinkler M, Ueland GA, Dennedy MC, Beuschlein F, Tabarin A, Fassnacht M, Ivovic M, Terzolo M, Kastelan D, Young WF Jr, Manolopoulos KN, Ambroziak U, Vassiliadi DA, Taylor AE, Sitch AJ, Nirantharakumar K, Arlt W; ENSAT EURINE-ACT Investigators*; ENSAT EURINE-ACT Investigators. Cardiometabolic Disease Burden and Steroid Excretion in Benign Adrenal Tumors : A Cross-Sectional Multicenter Study. Ann Intern Med. 2022 Mar;175(3):325-334. doi: 10.7326/M21-1737. Epub 2022 Jan 4. PMID 34978855
- [Background] Ebbehoj A, Li D, Kaur RJ, Zhang C, Singh S, Li T, Atkinson E, Achenbach S, Khosla S, Arlt W, Young WF, Rocca WA, Bancos I. Epidemiology of adrenal tumours in Olmsted County, Minnesota, USA: a population-based cohort study. Lancet Diabetes Endocrinol. 2020 Nov;8(11):894-902. doi: 10.1016/S2213-8587(20)30314-4. PMID 33065059
- [Background] Fassnacht M, Tsagarakis S, Terzolo M, Tabarin A, Sahdev A, Newell-Price J, Pelsma I, Marina L, Lorenz K, Bancos I, Arlt W, Dekkers OM. European Society of Endocrinology clinical practice guidelines on the management of adrenal incidentalomas, in collaboration with the European Network for the Study of Adrenal Tumors. Eur J Endocrinol. 2023 Jul 20;189(1):G1-G42. doi: 10.1093/ejendo/lvad066. PMID 37318239
- [Background] Kolanska K, Owecki M, Nikisch E, Sowinski J. High prevalence of obesity in patients with non-functioning adrenal incidentalomas. Neuro Endocrinol Lett. 2010;31(3):418-22. PMID 20588242
- [Background] Reimondo G, Castellano E, Grosso M, Priotto R, Puglisi S, Pia A, Pellegrino M, Borretta G, Terzolo M. Adrenal Incidentalomas are Tied to Increased Risk of Diabetes: Findings from a Prospective Study. J Clin Endocrinol Metab. 2020 Apr 1;105(4):dgz284. doi: 10.1210/clinem/dgz284. PMID 31900474
- [Background] Bovio S, Cataldi A, Reimondo G, Sperone P, Novello S, Berruti A, Borasio P, Fava C, Dogliotti L, Scagliotti GV, Angeli A, Terzolo M. Prevalence of adrenal incidentaloma in a contemporary computerized tomography series. J Endocrinol Invest. 2006 Apr;29(4):298-302. doi: 10.1007/BF03344099. PMID 16699294